CLINICAL TRIAL: NCT03932695
Title: Investigation of Milk Peptides on Postprandial Blood Glucose Profile: Randomized, Double-blind, Placebo-controlled, Cross-over Study With Different Dosages Followed by an Open-label Single Arm Phase to Estimate Long Term Effects
Brief Title: Investigation of Milk Peptides on Postprandial Blood Glucose Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredia S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTS1130/17
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: double blind cross over and open for the phase II of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: first phase of the study is RCT double blind placebo cross-over. The second phase is open during 6 weeks of supplementation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose Milk peptides (Active Comparator): 2800mg of whey protein hydrolysates single dose
  Interventions: Dietary Supplement: High Dose milk peptide
- Low dose Milk peptides (Active Comparator): 1400mg of whey protein hydrolysate Single dose and 6 weeks intervention
  Interventions: Dietary Supplement: Low dose milk peptide
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low dose milk peptide — what is the effect of milk peptides 1400mg on postprandial glycemia after a meal rich in carbohydrates (75g)
  Arms: Low dose Milk peptides
Dietary Supplement: High Dose milk peptide — what is the effect of milk peptides 2800mg on postprandial glycemia after a meal rich in carbohydrates (75g)
  Arms: High dose Milk peptides
Dietary Supplement: Placebo — what is the effect of placebo on postprandial glycemia after a meal rich in carbohydrates (75g)
  Arms: Placebo

SUMMARY:
Aim of the study is to investigate the effect of two different dosages of milk peptides on postprandial blood glucose profile in prediabetic subjects compared to placebo. This will be investigated in a cross-over double blind randomized placebo controlled study design. Additionally, long term effects on glucose status, insulin sensitivity and postprandial blood glucose profile will be investigated in a follow up 6-week open label phase with the low dose only.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with prediabetic HbA1c values between 5.7% - 6.4% and/or Fasting blood glucose ≥ 5.6 mmol/l (≥ 100 mg/dl) und < 7.0 mmol/l (< 125 mg/dl) (in venous plasma)
* Age: 30-70 years
* Body mass index 19-35 kg/m2
* Non-smoker
* Caucasian
* Availability and presence in the study unit for approx. 3.5 hours/ week for 3 times in a row with approx. 1 week of washout in between.
* Signed informed consent form
* No changes in food habits or physical activity 3 months prior to screening and during the study

Exclusion Criteria:

* Presence of disease or drug(s) influencing digestion and absorption of nutrients or bowel habits
* Intake of medications known to affect glucose tolerance, e.g., diabetic medication, steroids, protease inhibitors or antipsychotics
* Diagnosed Typ 2-Diabetics with medical treatment
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening)), which in the investigator's opinion would impact patient safety
* Severe liver, renal or cardiac disease
* Acute gastrointestinal diseases including diarrhea and/or vomiting within the last 2 weeks
* Known inflammatory and malignant gastrointestinal diseases (i.e. colitis ulcerosa, Morbus Crohn, celiac disease, malignant diseases e.g. colon-cancer, rectum cancer, pancreatitis)
* Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
* Major medical or surgical event requiring hospitalization within the previous 3 months
* Intake of antibiotics within 4 weeks before the test days
* Known alcohol abuse or drug abuse
* Pregnant or breast feeding women
* Known or suspected allergy to any component of the investigational product(s) (e.g. milk protein)
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study
* Subject unable to co-operate adequately
* Participation in a clinical study with an investigational product within one month before start of study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose-iAUC(0-180min) | day 1, day 8, day 15, day 57
  Area under the curve calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration

SECONDARY OUTCOMES:
Cmax | day 1, day 8, day 15, day 57
  Maximum blood glucose concentration
Max-Increase | day 1, day 8, day 15, day 57
  Cmax minus baseline value
Tmax | day 1, day 8, day 15, day 57
  Time to reach maximum blood glucose concentration
Tbaseline | day 1, day 8, day 15, day 57
  First time to reach baseline again after increase or decrease in blood glucose
AUC(0-180min): | day 1, day 8, day 15, day 57
  Total area under curve from 0 to 180 min for blood glucose concentration
Insulin-iAUC(0-180min) | day 1, day 8, day 15, day 57
  Area under the curve calculated as the incremental area under the Insulin response curve, ignoring the area beneath the fasting concentration
Cmax Baseline Insulin Max_increase Insulin | day 1, day 8, day 15, day 57
  Max_increase Insulin Cmax minus baseline insulin value
Tmax insulin | day 1, day 8, day 15, day 57
  time to reach maximum Insulin concentration
Fasting glucose, fasting insulin | Baseline and Day 57
HOMA index | Baseline and Day 57
  Parameters of insulin sensitivity:
HbA1c level | Baseline (V5) and Day 57 (after 6 weeks)
  HbA1c level after 6 weeks of supplementation
Matsuda index | Baseline and Day 57
  Insulin sensitivity
Quicki Index | Baseline and Day 57
  Insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Audrey BOULIER, MD, Principal Investigator — Ingredia S.A.
Locations (1):
- Biotesys, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No